CLINICAL TRIAL: NCT07362524
Title: Artificial Intelligence-assisted Optical Diagnosis for the Resect-and-discard Strategy in Clinical Practice in Non-academic Hospitals: a Randomized Controlled Study
Brief Title: AI-Assisted Real-Time Endoscopic Characterization of Diminutive Colorectal Polyps in Non-Academic Hospitals
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xiaobo Li, Chief physician, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: KY2024-080-A
Record Dates: First submitted 2025-09-27; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-10

CONDITIONS: Colorectal Polyps

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CADx assisted colonoscopy group (Experimental)
  Interventions: Device: AI-Assisted Real-time Endoscopic Diagnosis System
- Routine colonoscopy group (No Intervention): Endoscopists perform standard endoscopic diagnosis using conventional NBI-based NICE classification without AI assistance.

INTERVENTIONS:
Device: AI-Assisted Real-time Endoscopic Diagnosis System — CADx assists endoscopists in diagnosing colorectal diminutive polyps (<=5cm) during colonoscopy using narrow-band imaging (NBI). The system provides real-time prediction values of NICE classification for colorectal polyp. The intervention group receives AI-assisted diagnostic information displayed
  Arms: CADx assisted colonoscopy group

SUMMARY:
To validate the feasibility of promoting colorectal diminutive polyp "predict, resect, and discard" and "diagnose and leave" strategies for non-experts in general hospitals through CADx system.

DETAILED DESCRIPTION:
This study will: (1) develop and refine a deep learning model for optical diagnosis of diminutive colorectal polyps-predicting histologic type and the presence of advanced adenoma components-based on multicenter endoscopic videos; (2) conduct a randomized controlled study recruiting endoscopists from different regions and experience levels nationwide to evaluate, with or without access to the model's diagnostic output, the success rates of implementing the "resect and discard" and "diagnose and leave" strategies as well as identifying advanced adenoma components; and (3) carry out a prospective randomized controlled trial to assess the benefits of a real-time AI-assisted endoscopic system in facilitating endoscopists' implementation of the "resect and discard" and "diagnose and leave" strategies for diminutive colorectal polyps.

ELIGIBILITY:
Inclusion Criteria:

1. Agree to participate in this prospective randomized controlled study;
2. Age ≥18 years for colonoscopy;
3. At least one colorectal diminutive polyp (size <=5mm) found during examination;

Exclusion Criteria:

1. Already participating in other clinical trials, having signed informed consent and being in the follow-up period of other clinical trials;
2. Already participating in drug clinical trials and being in the washout period of experimental or control drugs;
3. History of drug or alcohol abuse or psychological disorders in the past five years;
4. Pregnant or lactating patients;
5. Known polyposis syndromes;
6. Patients with gastrointestinal bleeding;
7. Previous history of inflammatory bowel disease, colorectal cancer, or colorectal surgery;
8. Patients with contraindications to tissue biopsy;
9. Previous history of allergic reactions to bowel cleansing agent components;
10. Suffering from intestinal obstruction or perforation, toxic megacolon, heart failure (Grade III or IV), severe cardiovascular disease, severe liver failure, or renal insufficiency, etc.;
11. Patient's bowel preparation BBPS score <6 for this colonoscopy;
12. Researchers consider the patient unsuitable for trial participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 363 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-11-15 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
Agreement between optical- and histology-based post-polypectomy surveillance intervals according to United States Multi-Society Task Force (USMSTF) guidelines | 14 days
  The concordance between the follow-up intervals determined by endoscopists (integrating polyp pathology under high diagnostic confidence and pathology results under low diagnostic confidence) and the follow-up intervals based solely on pathological results, as recommended by the U.S. 2020 USMSTF consensus for post-polypectomy surveillance.
Negative Predictive Value for Diagnosing Neoplastic Lesions in Rectosigmoid Diminutive Polyps under High Confidence | 14 days

SECONDARY OUTCOMES:
Agreement between optical- and histology-based post-polypectomy surveillance intervals according to according to European Guidelines | 14 days
  The concordance between the follow-up intervals determined by endoscopists (integrating polyp pathology under high diagnostic confidence and pathology results under low diagnostic confidence) and the follow-up intervals based solely on pathological results, as recommended by the European ESGE 2020 consensus for post-polypectomy surveillance.
Agreement between optical- and histology-based post-polypectomy surveillance intervals according to Asia-Pacific Guidelines | 14 days
  The concordance between the follow-up intervals determined by endoscopists (integrating polyp pathology under high diagnostic confidence and pathology results under low diagnostic confidence) and the follow-up intervals based solely on pathological results, as recommended by the Asia-Pacific APWG 2022 consensus for post-polypectomy surveillance.
Agreement between optical- and histology-based post-polypectomy surveillance intervals according to Expert Consensus on Outpatient Management of Colorectal Polyps | 14 days
  The concordance between the follow-up intervals determined by endoscopists (integrating polyp pathology under high diagnostic confidence and pathology results under low diagnostic confidence) and the follow-up intervals based solely on pathological results, as recommended by the Expert Consensus on Outpatient Management of Colorectal Polyps (2025, Chengdu).
Diagnostic Accuracy, Sensitivity and Specificity for Diagnosing Neoplastic Lesions in Rectosigmoid Diminutive Polyps under High Diagnostic Confidence | 30 days
Diagnostic Accuracy, Sensitivity and Specificity for Diagnosing Neoplastic Lesions in Diminutive Polyps under High Diagnostic Confidence | 14 days
Diagnostic Accuracy of Endoscopists in Characterizing Colorectal Diminutive Polyps when assessed with High Diagnostic Confidence. | 14 days
Improvement in Endoscopists' Diagnostic Confidence with AI Assistance | 14 days
Improvement in Endoscopists' Diagnostic Accuracy in Characterizing Colorectal Diminutive Polyps with AI Assistance. | 14 days

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Nantong First People's Hospital, Nantong, Jiangsu
  - Wuxi Ninth People's Hospital, Wuxi, Jiangsu

IPD SHARING:
Plan to Share IPD: Yes